CLINICAL TRIAL: NCT04506749
Title: Clinical Trial to Evaluate the Efficacy of a Nutraceutical Versus Placebo in Reducing Cardiovascular Risk in Healthy Subjects
Brief Title: To Evaluate the Efficacy of a Nutraceutical in Reducing Cardiovascular Risk in Healthy Subjects
Acronym: JC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-00015
Record Dates: First submitted 2020-07-30; First posted 2020-08-10 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Consumption of antioxidant boiled ham, 100 grams daily to consume during the day.
  Consumption time: 8 weeks.
  Interventions: Dietary Supplement: Dietary supplement consumption
- control group Placebo (Placebo Comparator): Consumption of extra boiled ham, 100 grams daily to consume during the day. Consumption time: 8 weeks.
  Interventions: Dietary Supplement: Dietary supplement consumption

INTERVENTIONS:
Dietary Supplement: Dietary supplement consumption — The consumption time was 56 days. Consumed 100 grams daily to consume during the day.

SUMMARY:
Single-blind, double-blind, controlled, randomized clinical trial of two parallel branches depending on the product consumed (experimental product and placebo product) and single-center with the objective of evaluating the effect of the investigational product on cardiovascular risk reduction.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will make a total of two visits to the research laboratory and will carry out the tests established in the protocol. Subsequently, a statistical analysis will be performed with the variables measured in the study to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes (men or women) between 30 and 75 years of age, Caucasian.
* Present body mass index between 20 and 32 Kg / m2.
* Presenting fasting serum LDL-cholesterol levels equal to or greater than 110 mg / dL or total serum cholesterol equal to or greater than 180 mg / dL.
* Volunteers capable of understanding the clinical study and willing to grant written informed consent and to comply with study procedures and requirements.

Exclusion Criteria:

* Thyroid dysfunction, infections, or with any type of chronic disease (eg, autoimmune, inflammatory).
* Subjects who have suffered an ischemic-vascular event in the last months.
* Subjects in medication and / or nutraceutical treatment for hypertension, diabetes or hyperlipidemia (ex: statins).
* Subjects in treatment with drugs that due to their narrow therapeutic margin require monitoring of their plasma levels (digoxin, acenocoumarol, warfarin, etc ...).
* Subjects in treatment that affects body weight or appetite.
* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Subjects who are carrying out or intend to carry out any type of diet, low-calorie or not, during the study.
* Subjects who have donated a minimum of 0.5L of blood in the last month Vegetarian subjects.
* Subjects who have ingested omega 3 and / or 6 supplements in the last three months, (eg, fish oil, evening primrose oil, krill oil, or algae oil).
* Subjects under treatment with niacin or fibrates.
* Those subjects with alcohol abuse, or with excessive alcohol consumption (> 3 glasses of wine or beer / day) were excluded.
* Patients undergoing major surgery in the last 3 months.
* Smoking subjects or not, but in any case who have changed their nicotinic habits during their participation in the study.
* Participation in another clinical trial in the three months prior to the study.
* Lack of will or inability to comply with clinical trial procedures.
* Subjects whose condition did not make them eligible for the study according to the researcher's criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol | It is measured on an empty stomach, change after 56 days of consumption.
  Lipidic profile, measured in mg/dl
LDL - Cholesterol | It is measured on an empty stomach, change after 56 days of consumption.
  Lipidic profile, measured in mg/dl
HDL - Cholesterol | It is measured on an empty stomach, change after 56 days of consumption.
  Lipidic profile, measured in mg/dl
Triglycerides | It is measured on an empty stomach, change after 56 days of consumption.
  Lipidic profile, measured in mg/dl

SECONDARY OUTCOMES:
Assessing a change of blood pressure | Blood pressure measurements will be taken with a Holter monitor on two separate occasions and for 24 hours each day. Measurements were made at baseline and after 56 days of product consumption. Systolic and diastolic blood pressure will be measured
  blood pressure is measured with a holter
Blood glucose | It is measured on an empty stomach, before and after the consumption time (56 days).
  Glycidic analysis, measured in mg/dL
Glycosylated hemoglobin (HBA1c) | It is measured on an empty stomach, before and after the consumption time (56 days).
  Glycidic analysis, measured in %
malondialdehyde (MDA) | It is measured on an empty stomach, before and after the consumption time (56 days).
  oxidative damage, measured in ng/ml
Oxidized LDL | It is measured on an empty stomach, before and after the consumption time (56 days).
  oxidative damage, measured in pg/mL
Superoxide Dismutase (SOD) | It is measured on an empty stomach, before and after the consumption time (56 days).
  antioxidant defense, measured in pg/mL
Interleukin-6 (IL-6) | It is measured on an empty stomach, before and after the consumption time (56 days).
  Inflammation, measured in pg/mL
Proteins C Reactive (PCR) | It is measured on an empty stomach, before and after the consumption time (56 days).
  Inflammation, measured in mg/l
Fat mass | It is measured on an empty stomach, before and after the consumption time (56 days).
  Bioimpedance, in Kg.
Muscle mass | It is measured on an empty stomach, before and after the consumption time (56 days).
  Bioimpedance, in Kg.
Body mass index | It is measured on an empty stomach, before and after the consumption time (56 days).
  Bioimpedance, in Kg/m2.
Percentage of fat mass | It is measured on an empty stomach, before and after the consumption time (56 days).
  Bioimpedance, in %.
Control of dietary intake | A nutritional registry will be carried out. The nutritional intake of three days in two periods will be collected. One record at the beginning and another at the end, that is, six days.
  Diet source
Physical Activity Questionnaire | It is measured before and after the consumption time (56 days).
  Measured with the questionnaire Global Questionnaire on Physical Activity
Liver safety variables | It is measured on an empty stomach, before and after the consumption time (56 days).
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No